CLINICAL TRIAL: NCT06762951
Title: Pilates Mat Versus Segmental Control Exercises on Spinopelvic Angles in Patients with Chronic Non-Specific Low Back Pain
Brief Title: Pilates Mat Versus Segmental Control Exercises in Patients with Chronic Non-Specific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alyaa Mohamed Ahmed Mohamed Elgendy, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Spinopelvic Angels In CNSLBP
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Chronic Non-Specific Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group (A) (Experimental): Group (A): Twenty patients will receive Pilates mat exercise which consists of (single leg stretch + Pelvic press + Swimming + Opposite arm and leg reach + Side to side), 3 sets of 10 repetitions. And conventional physiotherapy treatment which consists of traditional physical therapy eg. (Back, hamstring, calf and hip flexors stretches, Abdominal curl-up exercise in supine, Back extensors exercise in prone, and Hip extensors exercises in prone along with ultrasound and Transcutaneous electrical nerve stimulation (TENS), two sessions per week for six weeks.
  Interventions: Other: Pilates mat exercices; Other: Traditional physical therapy
- Group (B) (Experimental): Group B: Twenty patients will receive Segmental control exercise which consists of (Segmental control over primary stabilizers, Exercises in closed chain, and Exercises in open chain) and conventional physiotherapy treatment which consists of traditional physical therapy eg. (Back, hamstring, calf and hip flexors stretches, Abdominal curl-up exercise in supine, Back extensors exercise in prone, and Hip extensors exercises in prone along with ultrasound and Transcutaneous electrical nerve stimulation (TENS), two sessions per week for six weeks
  Interventions: Other: Segmental control exercises; Other: Traditional physical therapy
- Group (C) (Active Comparator): Group C: Twenty patients will receive conventional physiotherapy treatment only which consists of traditional physical therapy eg. (Back, hamstring, calf and hip flexors stretches, Abdominal curl-up exercise in supine, Back extensors exercise in prone, and Hip extensors exercises in prone along with ultrasound and Transcutaneous electrical nerve stimulation (TENS), two sessions per week for six weeks.
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Pilates mat exercices — Pilates mat exercise which consists of (single leg stretch + Pelvic press + Swimming + Opposite arm and leg reach + Side to side), 3 sets of 10 repetitions.
  Arms: Group (A)
Other: Segmental control exercises — Segmental control exercise which consists of (Segmental control over primary stabilizers, Exercises in closed chain, and Exercises in open chain)
  Arms: Group (B)
Other: Traditional physical therapy — Traditional physical therapy eg. (Back, hamstring, calf and hip flexors stretches, Abdominal curl-up exercise in supine, Back extensors exercise in prone, and Hip extensors exercises in prone along with ultrasound and Transcutaneous electrical nerve stimulation (TENS)

SUMMARY:
This study sought to determine the effect of Pilates exercises versus segmental control exercises on spinopelvic angles, pain intensity, and functional disability in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is the most common musculoskeletal condition and constitutes a global public health problem. The majority of patients (up to 90%) are categorized as having nonspecific low back pain, which is described as symptoms lack of clear particular reasons, i.e., beginning of low back pain is not known. Many clinical guidelines and systematic reviews have recommended exercise therapy as one of the preferred treatments at decreasing pain and improving function in NSLBP. In the last decade, the Pilates method has become one of the most popular exercise programmes incorporated in clinical practice. Therapeutic exercises, specifically Segmental control exercises, decrease pain, reduce disability, improve quality of life, increase muscular endurance and strength, improve segmental stability, and reduce risk of injury. Studies have shown that both segmental control exercises and Pilate's exercises are effective in the management of pain and disability in individuals with Chronic LBP. However, it appears there is dearth of empirical data establishing which is more effective between the segmental control exercises and Pilates exercises on individuals with non-specific chronic low back pain. Thus, there exist certain gaps involving the two therapeutic techniques. Therefore, this study sought to determine the effect of Pilates exercises versus segmental control exercises on spinopelvic angles, pain intensity, and functional disability in patients with chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18 to 65 years. (Yentür et al., 2021)
* Both male and female gender will be included in the study. (Akhtar et al., 2017)
* Nonspecific, non-radicular (axial) chronic LBP diagnosis with hyperlordosis (LBP for at least three months). (Kızıltaş et al., 2022)
* Visual Analog Scale (VAS) score of 3 or higher. (Mannion et al., 2009)

Exclusion Criteria:

* Patients with acute attacks of LBP. (Caglayan et al.,2014)
* Pain referred from the lumbar to the lower extremities.
* Serious spinal disorder including malignancy, osteoporosis, ankylosing spondylitis, cauda equina compression, and infection.
* Fracture of vertebrae, and administered epidural injection. (Sarker et al., 2020)
* Pregnancy and feeding
* Structural abnormalities in the lumbar region
* Surgical history in the lumbar spine area
* Heart disease. (Kızıltaş et al., 2022)
* History of Vestibular dysfunction
* Regular Pilates/any other specific exercise program in the last 3 months. (Mehta et al.,2022)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Spinopelvic angels | 6 weeks
  Spinopelvic angles consists of (Sacral slope, lumber lordosis, pelvic incidence, and pelvic tilt) from the X-ray picture of the lateral view of the lumbosacral region by using CorelDraw graphic suits X7 software program. (Bhosale et al.2020)

SECONDARY OUTCOMES:
Pain intensity | 6 weeks
  Pain intensity by using a Visual analogue scale (VAS). (Begum, and Hossain 2019)
Functional disability | 6 weeks
  Functional disability by using the Oswestry disability questionnaire. (Koivunen et al., 2024)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Univercity, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Dimitrijevic V, Scepanovic T, Milankov V, Milankov M, Drid P. Effects of Corrective Exercises on Lumbar Lordotic Angle Correction: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2022 Apr 18;19(8):4906. doi: 10.3390/ijerph19084906. PMID 35457772
- [Background] Tamartash H, Bahrpeyma F. Evaluation of Lumbar Myofascial Release Effects on Lumbar Flexion Angle and Pelvic Inclination Angle in Patients with Non-Specific Low Back Pain. Int J Ther Massage Bodywork. 2022 Mar 2;15(1):15-22. doi: 10.3822/ijtmb.v15i1.709. eCollection 2022 Mar. PMID 35280247
- [Background] Koivunen K, Widbom-Kolhanen S, Pernaa K, Arokoski J, Saltychev M. Reliability and validity of Oswestry Disability Index among patients undergoing lumbar spinal surgery. BMC Surg. 2024 Jan 3;24(1):13. doi: 10.1186/s12893-023-02307-w. PMID 38172794
- [Background] Bhosale S, Pinto D, Srivastava S, Purohit S, Gautham S, Marathe N. Measurement of spinopelvic parameters in healthy adults of Indian origin - A cross sectional study. J Clin Orthop Trauma. 2020 Sep-Oct;11(5):883-888. doi: 10.1016/j.jcot.2019.07.013. Epub 2019 Jul 23. PMID 32879575
- [Background] Huang C, Hsieh YL, Chou LW, Wang JL, Chien A. Effects of pilates exercises on radiographic lumbo-pelvic alignment and range of motion in non-specific low back pain patients. J Bodyw Mov Ther. 2024 Apr;38:339-345. doi: 10.1016/j.jbmt.2023.10.004. Epub 2024 Feb 5. PMID 38763578